CLINICAL TRIAL: NCT03125798
Title: Comparison of LigaSure Technology to the Conventional Electrocoagulation in Video-assisted Thoracoscopic Surgery (VATS) Lobectomy Followed by Systemic Lymphadenectomy: A Prospective Randomized Controlled Study
Brief Title: Comparison of LigaSure to Conventional Electrocoagulation in Video-assisted Thoracoscopic Surgery Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wielkopolskie Centrum Pulmonologii i Torakochirurgii (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-17-ML-1
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer; Complication of Surgical Procedure
Keywords: video-assisted thoracic surgery; LigaSure; mediastinal lymph node dissection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LigaSure (Experimental): In this arm, LigaSure™ will be used for mediastinal lymph nodes dissection, according to standard surgical technique.
  Interventions: Device: LigaSure™
- Monopolar electrocautery (Active Comparator): In this arm, conventional monopolar electrocautery will be used for mediastinal lymph nodes dissection, according to standard surgical technique.
  Interventions: Device: Monopolar electrocautery

INTERVENTIONS:
Device: LigaSure™ — LigaSure™ is supposed to provide improved closure of lymphatic and blood vessels during mediastinal lymph nodes dissection.
  Arms: LigaSure
Device: Monopolar electrocautery — Monopolar electrocautery will be used according to the standard technique for the mediastinal lymph node dissection.
  Arms: Monopolar electrocautery

SUMMARY:
Surgical treatment of lung cancer consists of two elements: anatomical lung resection (segmentectomy, lobectomy or pneumonectomy) followed by mediastinal lymph node dissection (MLND). Since over last 15 years the growing rate of resection is performed by minimal invasive approach - video-assisted thoracoscopic surgery (VATS). The study is focused on the clinical and technical aspects of MLND during VATS lobectomy. The extension of lymph nodes resection is strictly specified. The main benefit of MLND for the patient is precise histopathological staging, which allows choosing the best therapeutic option of adjuvant therapy. MLND is related with potential minor and major complications (bleeding, increased volume of chest tube drainage, prolonged chest tube duration and hospital stay, chylothorax, left recurrent laryngeal nerve injury, injury of the bronchus, injury of the esophagus). The majority of complications are caused by thermal injury resulting from the use of heat-generating monopolar electrocautery that is commonly used during lymph nodes dissection. In addition, thermal energy generation in case of monopolar electrocautery may lead to systemic inflammatory response and increased surgical injury. High-energy sealing devices like LigaSure™ allow for dissection, coagulation and cutting with the single instrument. Compared to mechanical ligation techniques (vessel loops, clips) or monopolar electrocautery, LigaSure™ technology has been shown to reduce: intraoperative blood loss (in colorectal, gynecologic and urologic surgery), surgery time (in colorectal, gynecologic and urologic surgery), length of hospital stay (in gynecologic and urologic surgery). Investigators hypothesize that application of LigaSure™ in VATS anatomical resection may lead to diminished complications rate, lower systemic inflammatory response and shorter length of stay compared to monopolar electrocautery.

DETAILED DESCRIPTION:
Summary

Surgical treatment of lung cancer consists of two elements: anatomical lung resection (segmentectomy, lobectomy or pneumonectomy) followed by mediastinal lymph node sampling (MLNS) or mediastinal lymph node dissection (MLND). Since over last 15 years the growing rate of resection is performed by minimal invasive approach - video-assisted thoracoscopic surgery (VATS). This technique is used in at least 60% of patients with lung cancer operated on in the leading centers. The study project is focused on the clinical and technical aspects of MLNS/MLND during VATS lobectomy. Lymphadenectomy has to be performed obligatory in case of lung cancer resection. The extension of lymph nodes resection or sampling is strictly specified and should be the same independently from the surgical approach (thoracotomy or VATS). The main benefit of MLNS/MLND for the patient is precise histopathological staging, which allows choosing the best therapeutic option of adjuvant therapy. It was proved that MLND is superior to MLNS in its accuracy however the improvement of local control of the disease is not proved.

Mediastinal lymphadenectomy is related with potential minor and major complications. The risk of complications is low but in case of their occurrence hospital stay is usually significantly prolonged, quality of life decreases and additional surgery may be needed. In very small group of patients complications may lead to severe disability or death.

The most frequent complications related with MLND are:

1. Bleeding, sometimes requiring redo surgery;
2. Increased volume of chest tube drainage with prolonged chest tube duration and hospital stay;
3. Chylothorax;
4. Left recurrent laryngeal nerve injury;
5. Injury of the bronchus (especially of posterior part of right main bronchus during dissection of subcarinal lymph nodes);
6. Injury of the esophagus (dissection of subcarinal and paraesophageal lymph nodes).

The majority of the above mentioned complications are caused by thermal injury resulting from the use of heat-generating monopolar electrocautery that is commonly used during lymph nodes dissection. Bleeding or chylothorax are usually caused by incomplete blood or lymphatic vessels closure. Esophageal or bronchial wall injury can be caused by thermal injury followed by ischemia, necrosis and finally perforation. The diagnosis is frequently delayed. In addition, thermal energy generation in case of monopolar electrocautery may lead to systemic inflammatory response and increased surgical injury. Extent of surgical injury measured by acute phase proteins levels (c-reactive protein, alpha-1-antitrypsin, alpha-1-acid glycoprotein, haptoglobin) and interleukin levels was proved to be correlated to long-term results in patients with colorectal cancer.

Introduction of new high-energy sealing devices like LigaSure™ to clinical practice allows for dissection, coagulation and cutting with the single instrument. Compared to mechanical ligation techniques (vessel loops, clips) or monopolar electrocautery, LigaSure™ technology has been shown to significantly reduce:

* Operative blood loss in colorectal, gynecologic and urologic surgery
* Perioperative blood transfusions in gynecologic, urologic and general surgery
* Procedure time in colorectal, gynecologic and urologic surgery
* Length of hospital stay in gynecologic and urologic surgery.

There have been no randomized studies comparing the use of traditional electrocautery and LigaSure for lymphadenectomy during VATS resection due to non-small cell lung cancer.

Investigators hypothesize that application of LigaSure™ in VATS anatomical resection may lead to diminished complications rate, lower systemic inflammatory response and shorter length of stay compared to monopolar electrocautery.

Study design

Patients with early stage NSCLC who are routinely operated on by VATS will be randomized into two groups. First group called electro-VATS (Monopolar electrocautery) will be operated on with the use of traditional electrocautery and the second called liga-VATS (LigaSure) with the use of LigaSure. In the first group during the whole procedure (dissection of pulmonary ligament, mediastinal pleura and adhesions, as well as hilar dissection and lymphadenectomy) only traditional monopolar electrocautery will be used. In the liga-VASTS patients only LigaSure will be applied,no monopolar electrocautery will be used. The procedure of VATS lobectomy or segmentectomy will be performed in standardized fashion with separate stapling of hilar vessels and bronchus and lung parenchyma division. The hilar dissection and mediastinal lymphadenectomy will be performed using either monopolar electrocautery or LigaSure according to the randomization. The extent of lymphadenectomy will be the same in both groups and will include stations 2R,4R,7,8R,9R,10R,11R on the right side and stations 5,6,7,8L,9L,10L,11L on the left side. The number of removed lymph nodes will be counted. The extension of lymphadenectomy will be controlled and supervised by main investigator. Deep temperature inside the esophagus at the level approximately 2-3 cm below the carina will be measured during lymphadenectomy in order to assess the differences in the exposure of the surrounding tissues to the thermal energy generated by either LigaSure or electrocautery. The temperature measurement should in some part reflect the potential risk of thermal injury to the esophagus caused by different energy devices.

Investigators plan to enroll 200 patients, 100 patients in each group. Initial assessment will include age, gender, comorbidities (Charlson Comorbidity Index, CCI and Thoracic Revised Cardiac Risk Index, thRCRI scores) and pulmonary function tests. The following factors/parameters will be measured/compared in both groups: 24-hour, 48-hour and total volume of chest tube drainage, chest tube duration and hospital stay, rate of the prolonged air leak, rate of redo surgery due to bleeding, rate of postoperative complications related to the procedure, intraoperative blood loss and time of the surgery, local thermal effect, systemic inflammatory response after surgery.

Statistical analysis

The analyzed data will be presented as means, standard deviations, minimum and maximum values, medians, interquartile ranges (lower quartile, upper quartile) or percentage, as appropriate. Normality of the distribution will be tested with the Shapiro-Wilk's test, and the equality of variances will be checked with the Levene's test. For comparison of groups, unpaired t test or one-way ANOVA (for data which follow normal distribution and homogeneity of variances) or Welch test will be applied. In case data will not normally distributed nonparametric tests will be used - Mann-Whitney U test or the Kruskal-Wallis test with the Dunn's post-hoc test. Categorical data will be analyzed with the χ2 test or the Fisher-Freeman-Halton test. The relationship between variables will be analyzed with the Pearson's linear correlation coefficient or the Spearman's rank correlation coefficient or (and) by multivariate linear regression. All the results will be considered significant at p<0.05. Statistical analyses will be performed with statistical packages: STATISTICA 10.0 PL (StatSoft. Inc.) or StatXact 9.0 (CytelStudio) software.

ELIGIBILITY:
Inclusion Criteria:

* Surgery performed by Video-Assisted Thoracic Surgery technique (VATS).
* Mediastinal Lymph Node Dissection performed due to the European Society of Thoracic Surgeons
* Patients must be informed and must sign and give written informed consent.

Exclusion Criteria:

* Preoperative radiotherapy.
* Preoperative chemotherapy.
* Mediastinoscopy or other surgical procedures of mediastinum prior to the present surgery.
* Chest surgery on the side to be operated.
* Conversion from VATS to thoracotomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Piwkowski, Prof, Principal Investigator — Wielkopolskie Centrum Pulmonologii i Torakochirurgii
Locations (1):
- Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- [Background] Lesser TG, Wolfram F, Boltze C. Sealing of pulmonary arteries with LigaSure: in vivo and ex vivo examinations. J Thorac Cardiovasc Surg. 2013 Jun;145(6):1525-8. doi: 10.1016/j.jtcvs.2012.11.009. Epub 2012 Dec 8. PMID 23228409
- [Background] Piccinni G, Pasculli A, D'Ambrosio E, Gurrado A, Lissidini G, Testini M. Retrospective comparison of Traditional vs. LigaSure impact dissection during pancreatoduodenectomy: how to save money by using an expensive device. Surg Technol Int. 2013 Sep;23:88-93. PMID 24081851
- [Background] Lee WJ, Chen TC, Lai IR, Wang W, Huang MT. Randomized clinical trial of Ligasure versus conventional surgery for extended gastric cancer resection. Br J Surg. 2003 Dec;90(12):1493-6. doi: 10.1002/bjs.4362. PMID 14648726
- [Background] Bertolaccini L, Viti A, Cavallo A, Terzi A. Results of Li-Tho trial: a prospective randomized study on effectiveness of LigaSure(R) in lung resections. Eur J Cardiothorac Surg. 2014 Apr;45(4):693-8; discussion 698. doi: 10.1093/ejcts/ezt445. Epub 2013 Sep 12. PMID 24031044
- [Background] Kuroda H, Dejima H, Mizumo T, Sakakura N, Sakao Y. A new LigaSure technique for the formation of segmental plane by intravenous indocyanine green fluorescence during thoracoscopic anatomical segmentectomy. J Thorac Dis. 2016 Jun;8(6):1210-6. doi: 10.21037/jtd.2016.04.61. PMID 27293839
- [Derived] Gabryel P, Roszak M, Skrzypczak P, Gabryel A, Zielinska D, Sielewicz M, Campisi A, Kasprzyk M, Piwkowski C. Identification of Factors Related to the Quality of Lymphadenectomy for Lung Cancer: Secondary Analysis of Prospective Randomized Trial Data. J Clin Med. 2023 May 31;12(11):3780. doi: 10.3390/jcm12113780. PMID 37297976
- [Derived] Gabryel P, Kasprzyk M, Roszak M, Campisi A, Smolinski S, Zielinski P, Piwkowski C. Comparison of the LigaSure bipolar vessel sealer to monopolar electrocoagulation for thoracoscopic lobectomy and lymphadenectomy: a prospective randomized controlled trial. Surg Endosc. 2023 Jun;37(6):4449-4457. doi: 10.1007/s00464-023-09892-0. Epub 2023 Feb 15. PMID 36792782

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LigaSure | Monopolar Electrocautery
Started | 109 | 107
Completed | 100 | 100
Not Completed | 9 | 7
Not completed — Lack of electrosurgical device in the operating room | 2 | 0
Not completed — Conversion to thoracotomy | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LigaSure | Monopolar Electrocautery | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.4) | 66.4 (7.3) | 66.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 58 | 58 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 100 | 100 | 200
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Chest Drainage Volume up to Chest Drain Removal, Average 3 Days.
Description: Measurement of the postoperative volume of fluid drained in milliliters, measured up to chest drain removal, average 3 days.
Time Frame: Total postoperative chest drainage volume
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | LigaSure | Monopolar Electrocautery
Number analyzed (Participants) | 100 | 100
ml | 550 [335 to 905] | 580 [352 to 950]

2. Secondary Outcome: Acute Phase Proteins Levels.
Description: Change in C-reactive protein (CRP) level, calculated as the difference between CRP values [mg/L] at 72 hours after surgery and 24 hours before surgery
Time Frame: 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | LigaSure | Monopolar Electrocautery
Number analyzed (Participants) | 98 | 95
mg/L | 68.5 [37.9 to 116.0] | 69.2 [44.8 to 107.4]

3. Secondary Outcome: Local Temperature.
Description: Change in the intraesophageal temperature at the level of the subcarinal lymph nodes, calculated as the difference between the highest temperature during subcarinal nodes dissection and the temperature before subcarinal nodes dissection
Time Frame: During mediastinal lymph nodes dissection (during surgery)
Measure: Median (Inter-Quartile Range); unit: degree Celcius
Arm/Group | LigaSure | Monopolar Electrocautery
Number analyzed (Participants) | 87 | 88
degree Celcius | -0.1 [-0.2 to 0.1] | -0.1 [-0.2 to 0.1]

ADVERSE EVENTS:
Time Frame: Data were collected from the beginning of the intervention (first use of the LigaSure device or monopolar device during surgery) until hospital discharge, an average of 1 week"
Arm/Group | LigaSure | Monopolar Electrocautery
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 24/100 | 22/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LigaSure (N=100) | Monopolar Electrocautery (N=100)
Prolonged air leak (Surgical and medical procedures) | 10 | 12
Residual air space (Surgical and medical procedures) | 8 | 7
Atrial fibrillation (Surgical and medical procedures) | 6 | 3

LIMITATIONS AND CAVEATS:
It was not possible to conceal the type of intervention - dissection with LigaSure versus monopolar device - from the surgeons who performed the operations. Methodological limitations may have resulted in the non-detection of the differences in intra-esophageal temperature and energy-dissipation-related complications between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03125798/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03125798/SAP_001.pdf